CLINICAL TRIAL: NCT05982665
Title: Effect of Inhaled Molecular Hydrogen on Recovery Process After Downhill Walking on the Treadmill. A Randomized, Double-blind, Placebo-controlled Crossover Study
Brief Title: Effect of Inhaled Molecular Hydrogen on Recovery Process After Downhill Walking on the Treadmill
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palacky University (Other)
Responsible Party: Principal Investigator, Jakub Krejci, Assistant professor, Palacky University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: FTK_2023_12
Record Dates: First submitted 2023-07-30; First posted 2023-08-08 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Muscle Soreness; Muscle Fatigue; Oxidative Stress; Inflammation
MeSH Terms: conditions — Myalgia; Inflammation | interventions — Hydrogen

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Hydrogen and placebo generators indistinguishable to the human senses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Molecular hydrogen (Experimental): Molecular hydrogen inhalation for 60 min at 48 h, 24 h, and 60 min pre-exercise and for 30 min post-exercise and 24 h post exercise.
  Interventions: Other: Molecular hydrogen
- Placebo (Placebo Comparator): Placebo inhalation for 60 min at 48 h, 24 h, and 60 min pre-exercise and for 30 min post-exercise and 24 h post exercise.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Molecular hydrogen — Hydrogen gas, purity >99.9%, flow rate 300 ml/min.
  Other Names: i300 Hydrogen Generator, H2 World Health & Beauty Company, Ostrava, Czech Republic
  Arms: Molecular hydrogen
Other: Placebo — Ambient air, flow rate 300 ml/min.
  Other Names: i300 Placebo Generator, H2 World Health & Beauty Company, Ostrava, Czech Republic
  Arms: Placebo

SUMMARY:
This study assesses the effect of molecular hydrogen inhalation in healthy males on muscle soreness, fatigue, oxidative stress, and inflammation following eccentric muscle contraction during downhill walking on the treadmill.

DETAILED DESCRIPTION:
The main aim of this randomized, double-blind, placebo-controlled crossover study is to assess the effect of molecular hydrogen inhalation on recovery after downhill walking with an additional load of 15% of body mass on the treadmill with a negative slope of -15% at a speed of 6.5 km/h for 90 min. The study includes 12 participants, healthy males aged 20-35 years. The study consists of two experimental sessions, one using molecular hydrogen inhalation and the other using placebo inhalation. Randomization is performed using a computer random generator. Molecular hydrogen is colourless, odourless, and tasteless, so it cannot be distinguished from placebo by the human senses. The washout period between sessions is set at four weeks. One week before each session, participants are asked to follow diet and physical activity rules. Variables measured during the 48 h recovery are as follow: creatine kinase level, perceived muscle soreness, reactive strength index, malondialdehydes level, and interleukin-6 level. The following variables are also measured during exercise: heart rate, ventilation and gas exchange, and blood lactate level. Analysis of variance for repeated measures and Fisher's post hoc tests are used for statistical analysis. The significance level is set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Free of major diseases.
* Completed questionnaire Sudden Cardiovascular Death in Sport: Lausanne Recommendations.
* Signed informed consent.

Exclusion Criteria:

* Acute conditions contraindicating laboratory testing of sports performance.
* Hypertension.
* Dyslipoproteinaemia.
* Cardiorespiratory disease.
* Pharmacotherapy affecting heart rate.
* Musculoskeletal problems.

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2023-08-14 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2023-11-29 (Actual)

PRIMARY OUTCOMES:
Creatine kinase | Change between values before and after 4 weeks of crossover.
  The level of creatine kinase is measured from a venous blood sample taken by a healthcare specialist. Samples are collected in 2.7 ml citrate vacuum tubes. Samples are immediately centrifuged at 1000 g for 15 min and then divided into 0.5 ml cryotubes and frozen at -80 °C. Samples are taken pre-exercise (baseline), post-exercise, and 2 h, 24 h and 48 h post-exercise. Creatine kinase is determined by ELISA method according to the manufacturer's instructions.
Perceived muscle soreness | Change between values before and after 4 weeks of crossover.
  A visual analogue scale is used to subjectively assess lower limb muscle soreness. The visual analogue scale is represented by a 100 mm line marked 0 - no pain and 100 - worst imaginable pain. The subject is instructed to mark a point on the line corresponding to their perceived muscle soreness. Muscle soreness is assessed pre-exercise (baseline), post-exercise, and 2 h, 24 h and 48 h post-exercise.

SECONDARY OUTCOMES:
Reactive strength index | Change between values before and after 4 weeks of crossover.
  Reactive strength index is determined in 5 maximum hop test on AMTI OR6-7-1000 force platform (Advanced Mechanical Technology, Watertown, USA). Each subject is instructed to maximize the jump height and minimize the ground contact time. Reactive strength index is measured pre-exercise (baseline), post-exercise, and 2 h, 24 h and 48 h post-exercise.
Malondialdehydes | Change between values before and after 4 weeks of crossover.
  The level of malondialdehydes is measured from a venous blood sample taken by a healthcare specialist. Samples are collected in 2.7 ml citrate vacuum tubes. Samples are immediately centrifuged at 1000 g for 15 min and then divided into 0.5 ml cryotubes and frozen at -80 °C. Samples are taken pre-exercise (baseline), post-exercise, and 2 h post-exercise. Malondialdehydes are determined using TBARS assay kit according to the manufacturer's instructions.
Interleukin-6 | Change between values before and after 4 weeks of crossover.
  The level of Interleukin-6 is measured from a venous blood sample taken by a healthcare specialist. Samples are collected in 2.7 ml citrate vacuum tubes. Samples are immediately centrifuged at 1000 g for 15 min and then divided into 0.5 ml cryotubes and frozen at -80 °C. Samples are taken pre-exercise (baseline), post-exercise, and 2 h post-exercise. Interleukin-6 is determined by ELISA method according to the manufacturer's instructions.

OTHER OUTCOMES:
Heart rate | Change between values before and after 4 weeks of crossover.
  Heart rate during the 90 min exercise is continuously recorded by Polar V800 heart rate monitor (Polar, Kempele, Finland).
Ventilation | Change between values before and after 4 weeks of crossover.
  Ventilation (air flow into and out of the lungs expressed in L/min) is measured with Ergostik analyser (Geratherm Respiratory, Bad Kissinger, Germany) breath by breath during the exercise and averaged over 5 min windows for subsequent analysis.
Oxygen uptake | Change between values before and after 4 weeks of crossover.
  Oxygen uptake is measured with Ergostik analyser (Geratherm Respiratory, Bad Kissinger, Germany) breath by breath during the exercise and averaged over 5 min windows for subsequent analysis.
Blood lactate | Change between values before and after 4 weeks of crossover.
  The level of blood lactate is measured from the fingertip blood sample using Lactate Scout+ analyser (EKF Diagnostics, Cardiff, UK) pre-exercise (baseline) and at specified time points (30, 60, and 90 min) during the exercise.
Rating of perceived exertion | Change between values before and after 4 weeks of crossover.
  Subjects are asked to subjectively rate their perceived exertion at specified time points (30, 60, and 90 min) during the exercise. The Borg's scale 6 (no exertion at all) and 20 (maximal exertion) is used.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Jarmar, Mgr, Principal Investigator — Palacky University, Faculty of Physical Culture
Locations (1):
- Palacky University, Faculty of Physical Culture, Olomouc, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Anonymised raw data will be made available.
Time Frame: The data will be available once the results are published in a scientific journal.
Access Criteria: For everybody.